CLINICAL TRIAL: NCT05200663
Title: Comparison of the Efficacy of the Tamoxifen and Tamoxifen With Antioxidants on Semen Quality of Infertile Male With Abnormal Semen Parameters.
Brief Title: Efficacy Comparison of Tamoxifen and Tamoxifen With Antioxidants on Semen Quality of Male With Idiopathic Infertility
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sharif Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMDC/SMRC/213-21/2021
Record Dates: First submitted 2021-11-24; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Oligoasthenoteratozoospermia; Male Infertility
Keywords: Tamoxifen citerate; Anti oxidants
MeSH Terms: conditions — Oligospermia; Infertility, Male | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: 110 patients are recruited into two groups .55 patients in group A will be given tamoxifen 10 mg twice a day and 55 patients in group B will be given tamoxifen 10 mg twice a day and vit E 400mg once a day.
Who Masked: Participant
Masking Description: It is single blinded study in which 110 patients are recruited into two groups .Randomization will be done by lottery method to divide the patients into group A & group B. 55 patients in group A will be given tamoxifen 10 mg twice a day and 55 patients in group B will be given tamoxifen 10 mg twice a day and vit E 400mg once a day. Only researcher will be knowing that which treatment will be giving to which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Tamoxifen" (Experimental): Group A patients will receive tab tamoxifen 10 mg twice a day for total of six months.
  Interventions: Drug: Tab Tamoxifen 10 mg
- "Tamoxifen and Antioxidant" (Active Comparator): Group B patients will receive tab tamoxifen 10 mg twice a day and cap. vit E 400mg once a day for total of six months.
  Interventions: Drug: Tab Tamoxifen 10mg,Cap vitamin E 400mg

INTERVENTIONS:
Drug: Tab Tamoxifen 10 mg — Tablet tamoxifen 10mg twice a day for 6 months.
  Other Names: Group A
  Arms: "Tamoxifen"
Drug: Tab Tamoxifen 10mg,Cap vitamin E 400mg — Tab tamoxifen 10 mg is given twice a day and cap vit E 400mg is given once a day for 6 months
  Other Names: Group B
  Arms: "Tamoxifen and Antioxidant"

SUMMARY:
Objective of the study is to compare the efficacy of tamoxifen alone & tamoxifen with antioxidant on semen quality of infertile male with abnormal parameters (sperm count, motility, vitality, morphology) .Infertility is defines as inability to conceive after one year of unprotected and regular intercourse. Infertility is the most important issue in the married couples and is one of the major clinical problem affecting people medically and psychologically .It affects about 5.8 to 44.2 % couples in the developing countries. Male infertility contributes to about 50% of the overall infertility. Antiestrogens are considered as one of the old and most commonly prescribed treatment of idiopathic infertility.Many studies has shown that it improves idiopathic oligozoospermia, count, motility and vitality. Spermatozoa are also prone to oxidative damage.

Men who have high reactive oxygen species(ROS) may have lower fertility potential as compared to men with low ROS. High levels of ROS in semen have been correlated with reduced sperm motility and damage to sperm nuclear DNA. High levels of cytokines in the semen is correlated with sperm injury like cell membrane lipid peroxidation in the presence of raised IL-6 .Antioxidents are the most important form of protection for spermatozoa against ROS. So oral antioxidents are commonly prescribed to males with idiopathic abnormal semen parameters and infertility to reduce the oxidative stress and improves infertility.

It is a single blinded randomized control trial to be conducted in Sharif Medical and Dental college, Lahore with sampling technique of probability randomized consecutive sampling technique. 110 male patients with idiopathic male infertility and abnormal semen parameters will be recruited . Pre treatment semen analysis and LH, FSH and serum testosterone will be done. 55 patients will be given tamoxifen alone ad 55 patients will be given tamoxifen with antioxidant. Then at the interval of 3 and 6 months after treatment , semen analysis and hormonal profile will be repeated. Pre-treatment and post treatment semen parameters will be compared using paired sample t-test. P-value < 0.05 will be taken as significant.

DETAILED DESCRIPTION:
Infertility is considered as the most important issue among the married couples and it represents major clinical problems affecting people not just medically but also psychologically .

Infertility affects about 5-8% of couple in developed countries and 5.8 - 44.2% in developing nations. In Pakistan incidence of oligozoospermia is around 21 percent and 12.32 % of patients presents with azoospermia (2). Male infertility contributes to about 50% of the cases of infertility . Cause of male infertility with abnormal semen parameters remains unknown in about 25% of men Men with idiopathic infertility may receive number of empirical therapies by clinicians. Commonly prescribed medications include hormonal medications such as follicular stimulating hormone (FSH), androgens like testosterone and mesterolone, antiestrogens ( tamoxifine, clomiphene citrate) , antioxidents like vitamin E, glutathione and sperm vitalizer such as L-carnitine ,coQ10.

Antiestrogens are considered to be one of the oldest and most commonly prescribed treatment for the idiopathic male infertility. Antiestrogen given for 6-9 months reported to have pregnancy rate of 20-40% . According to WHO tamoxifen citerate is the first line treatment for idiopathic ologozoospermia . Previously tamoxifen citrate was given as the empirical treatment for oligozoospermia and later it was found that after the use of 3-6 months it improves sperm count, motility and viability . The exact mechanism by which tamoxifen increase sperm parameters is not known , however it is found that it has stimulatory action on gonadotrophin secretion and directly effects leydig cell function . Tamoxifen is also known for the treatment of breast cancer worldwide.

Oxidative stress has been widely studied previously as one of the cause of the male infertility. Like other aerobic cells , spermatozoa are also prone to the oxidative damage because they have large polyunsaturated fat content in their membrane. Men who have high reactive oxygen species(ROS) may have lower fertility potential as compared to men with low ROS. High levels of ROS in semen have been correlated with reduced sperm motility and damage to sperm nuclear DNA. High levels of cytokines in the semen is correlated with sperm injury like cell membrane lipid peroxidation in the presence of raised IL-6 . Interferone gamma and TNF alpha have shown to decrease the motility of spermatozoa. This is commonly present in genitourinary infections and inflammation in which oxidative mechanism can leads to oxidative stress . Antioxidents are the most important form of protection for spermatozoa against ROS. So oral antioxidents are commonly prescribed to males with idiopathic abnormal semen parameters and infertility to reduce the oxidative stress and improves infertility.

Though assisted reproductive techniques are being widely offered to infertile couples, however before referring the patients for these expensive treatment options , relatively economical and practical methods should be considered first.

This study has been designed to determine the improvement of semen quality of infertile male with abnormal parameters after treatment with tamoxifen & tamoxifen with antioxidants thus the chances of conception and pregnancy rates are expected to be improved.

OBJECTIVE:

To compare the efficacy of tamoxifen alone & tamoxifen with antioxidant on semen quality of infertile male with abnormal parameters (sperm count, motility, vitality, morphology) .

OPERATIONAL DEFINITIONS:

Infertility: Inability to conceive after one year of unprotected and regular intercourse.

Abnormal Semen parameters:

Oligospermia: A sperm count of less than 15 million/ml .

Azoospermia: Absence of spermatozoa in the semen. Asthenozoospermia: reduced sperm motility. Teratozoospermia: presence of spermatozoa with abnormal morphology Asthenoteratozoospermia: Abnormal sperm motility and morphology

MATERIALS AND METHODS:

Study Design: Single Blind Randomized Controlled Trial Setting: Department of Obstetrics and Gynecology, Sharif Medical City, Lahore for 1 years.

Sampling Technique: Probability Randomized Consecutive Sampling Technique.

SAMPLE SELECTION:

Sample Size: A sample size of 110 (55in each group) with 95% confidence interval at 5% level of significance.

DATA COLLECTION PROCEDURE:

After approval of proposed synopsis from the ethical review board, infertile males with abnormal semen parameters will be included in the study after written informed consent. Randomization will be done by lottery method to divide the patients into group A & group B.

In group A: Tab. Tamoxifen 10 mg ,per oral twice daily will be given for six months.

In group B: Tab. Tamoxifen 10mg twice a day and Cap Evion 400mg once a day will be given for six months.

Semen analysis will be performed, according to the WHO criteria 20101, on all the patients for measurement of semen parameters ( volume, sperm concentration, total sperm number, motility & morphology) All samples will be collected in a private room at the laboratory in Sharif medical city, wide-mouth container kept at body temperature, after abstaining from any sexual activity for no less than 3 and no more than 7 days. Masturbation will be used as the method of sample production, without the use of any lubricants, after washing and drying both the hands and the penis. The sample is then incubated at 37 ºC till liquefaction is complete.

Semen volume will be measured in a graduated cylinder, whereas, sperm count and morphology will be assessed by microscopy. Sperms appearing within a square on the grid pattern will be counted to determine the sperm count.

Hormonal profile such as Serum FSH, serum LH and Serum Testosterone of all patients will also be analyzed before starting the treatment. Semen samples and hormonal profile will be analyzed pre-treatment and at interval of three months and six months after treatment. All the research data will be taken on a pre-designed Performa.

DATA ANALYSIS:

Data analysis will be done using SPSS v 23. Quantitative variables such as age, sperm count, motility, and vitality concentration will be analyzed and mean and standard deviation will be calculated. Independent sample test will be used to compare quantitative variables between the groups. While pre-treatment and post treatment semen parameters will be compared using paired sample t-test. P-value < 0.05 will be taken as significant. Bias will be reduced by using the same laboratory for all tests. Data, will be stratified for age, BMI, smoking ,alcohol drinking, baseline sperm parameters (sperm count, concentration , motility, vitality) and hormone assays (follicular stimulating hormone (FSH), luteinizing hormone(LH) and testosterone).

ELIGIBILITY:
Inclusion Criteria:

- All infertile male with idiopathic infertility and abnormal semen analysis.

Exclusion Criteria:

* 1. Leukocytospermia i.e. significant WBCs seen in the semen, 2. Severe oligospermia (sperm count <5 million per ml),

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All infertile males fulfilling the inclusion criteria.
Enrollment: 110 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Semen Volume | at 3 months posttreatment
  Semen Volume measured in ml.
Semen Volume | at 6 months posttreatment
  Semen Volume measured in ml.
Total sperm Count | 3 months posttreatment
  Total Sperm No.(x106)
Total sperm Count | 6 months posttreatment
  Total Sperm No.(x106):
Sperm concentration | 3 months posttreatment
  Sperm Conc. (x106)/ ejeculate:
Sperm concentration | 6 months posttreatment
  Sperm Conc. (x106)/ ejeculate:
Progressive motility | 3 months posttreatment.
  Progressive motility in (Percentage %):
Progressive motility | 6 months posttreatment
  Progressive motility (Percentage %):
Sperm Morphology: | 3 months posttreatment
  Sperm Morphology: Percentage %
Sperm Morphology: | 6 months posttreatment
  Sperm Morphology: Percentage %
Vitality | 3 months posttreatment
  Vitality (live spermatozoa in percentage%
Vitality | 6 months posttreatment
  Vitality (live spermatozoa) in percentage%
Leutinizing hormone | 3 months posttreatment
  Leutinizing hormone (LH) measured in mU/ml
Leutinizing hormone | 6 months posttreatment
  Leutinizing hormone (LH) measured in mU/ml
Follicular stimulating hormone | 3 months posttreatment.
  Follicular stimulating hormone (LH) measured in mU/ml
  Follicular stimulating hormone (FSH) measured in mU/ml
Follicular stimulating hormone | 6 months posttreatment.
  Follicular stimulating hormone (LH) measured in mU/ml
  Follicular stimulating hormone (FSH) measured in mU/ml
Serum Testosterone | 3 months posttreatment.
  Serum Testosterone measured in ng/dl
Serum Testosterone | 6 months posttreatment.
  Serum Testosterone measured in ng/dl

CONTACTS AND LOCATIONS:
Overall Officials: Anees Fatima, MBBS,FCPS, Principal Investigator — Sharif Medical And Dental College
Locations (1):
- Sharif Medical And Dental College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meng Q, Ren A, Zhang L, Liu J, Li Z, Yang Y, Li R, Ma L. Incidence of infertility and risk factors of impaired fecundity among newly married couples in a Chinese population. Reprod Biomed Online. 2015 Jan;30(1):92-100. doi: 10.1016/j.rbmo.2014.10.002. Epub 2014 Oct 13. PMID 25456165
- [Result] Butt F, Akram N. Semen analysis parameters: experiences and insight into male infertility at a tertiary care hospital in Punjab. J Pak Med Assoc. 2013 May;63(5):558-62. PMID 23757979
- [Result] Safarinejad MR. The effect of coenzyme Q(1)(0) supplementation on partner pregnancy rate in infertile men with idiopathic oligoasthenoteratozoospermia: an open-label prospective study. Int Urol Nephrol. 2012 Jun;44(3):689-700. doi: 10.1007/s11255-011-0081-0. Epub 2011 Nov 13. PMID 22081410
- [Result] Siddiq FM, Sigman M. A new look at the medical management of infertility. Urol Clin North Am. 2002 Nov;29(4):949-63. doi: 10.1016/s0094-0143(02)00085-x. PMID 12516764
- [Result] 5. Iacono F, Prezioso D, Ruffo A et al. Treating idiopathic male infertility with a combination of tamoxifen citrate and a natural compost of antioxidant and androgen mimetic action. J Steroid Hormone Sci. 2013;S5: 1-6.
- [Result] Kadioglu TC. Oral tamoxifen citrate treatment is more effective in normogonadotropic patients who have follicle-stimulating hormone levels within the lower half of normal. Int Urol Nephrol. 2009 Dec;41(4):773-6. doi: 10.1007/s11255-009-9568-3. Epub 2009 Apr 21. PMID 19381855
- [Result] Adamopoulos DA. Medical treatment of idiopathic oligozoospermia and male factor subfertility. Asian J Androl. 2000 Mar;2(1):25-32. PMID 11228933
- [Result] Nada EA, El Taieb MA, Ibrahim HM, Al Saied AE. Efficacy of tamoxifen and l-carnitine on sperm ultrastructure and seminal oxidative stress in patients with idiopathic oligoasthenoteratozoospermia. Andrologia. 2015 Sep;47(7):801-10. doi: 10.1111/and.12333. Epub 2014 Oct 2. PMID 25274200
- [Result] Sharma RK, Agarwal A. Role of reactive oxygen species in male infertility. Urology. 1996 Dec;48(6):835-50. doi: 10.1016/s0090-4295(96)00313-5. PMID 8973665